CLINICAL TRIAL: NCT02569580
Title: Clinical Trial of Anti-Lice Treatment Using the Medical Device "No More" Which is Designed to Kill Lice and Lice Eggs on the Head.
Brief Title: Effectiveness of "No More" Anti-lice Medical Device to Kill Lice and Lice Eggs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pharmayeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0022-14-LND
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Lice
Keywords: anti-lice treatment
MeSH Terms: conditions — Lice Infestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Topically — use the "No More" medical device as anti lice treatment

SUMMARY:
The purpose of this study is to determine effectiveness of an Anti-lice treatment using the medical device "No More" which is designed to kill lice and lice eggs on the head.

DETAILED DESCRIPTION:
The Clinical Trial Protocol include 2 visits

First Visit: Explanation and signing of consent forms. Diagnosis: Prof. Shemer will check if the patients have sufficient living lice or lice eggs and if so they will be scheduled to receive treatment.

Second Visit: -Spread the "No More" on the head of the boy or girl on dry hair.

* After five minutes comb with an adequately thick comb and the eggs will fall out easily with the pulling of the comb.
* Wash the hair.
* Combing the hair again with a thick comb for five minutes and/or 20 combings; Checking if the head is free of eggs and lice via a visual inspection by the head researcher.

Outcome

1. If there are no live eggs and/or lice then the patient has completed treatment - and the research. (This outcome is defined as successful treatment.)
2. If there are eggs only then the patient is scheduled for a third visit after seven days (+/- one day).
3. If live lice are found this outcome is defined as failure and the patient will not be scheduled for an additional visit

Third Visit:

After seven days (+/- one day) Professor Shemer will conduct a visual inspection for lice and lice eggs. Combing with a thick comb for five minutes and/or 20 combings and if there are live lice or lice eggs

Treatment Success:

No eggs and no lice immediately with the end of the treatment (second visit). No lice or live lice eggs after seven days (+/- one day).

Number of Participants: Up to 80 participants when at least 50 participants complete the treatment.

Age Range: 3-18 years

ELIGIBILITY:
Inclusion Criteria:

Patients that are suffering from lice and lice eggs that agree to refrain from any other treatment or salve designed for the treatment of lice and/or lice eggs throughout the course of the research study.

Patients that orally and in writing express their agreement to participate in the study - Consent in writing will be provided by two parents; Oral consent will be provided by the participants themselves.

Exclusion Criteria:

Pregnant or nursing women.

Patients lacking the faculties for proper judgment.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
No live lice eggs and/or live lice | 1 day from second visit

CONTACTS AND LOCATIONS:
Overall Officials: Ben Berger, Study Director — Prof. Avner Shemer clinic
Locations (1):
- Prof. Avner Shemer clinic, Netanya, Israel